CLINICAL TRIAL: NCT04634188
Title: Role and Value of Inflammatory Markers in Brain Tumors : A Case Controlled Study
Status: Completed | Type: Observational
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, Ridha Dharmajaya, Prof. Dr., Universitas Sumatera Utara
Other Study IDs: Universitas Sumatera Utara
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Brain Tumor
Keywords: Brain Tumor, Inflammation, Procalcitonin, CRP, NLR
MeSH Terms: conditions — Brain Neoplasms; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Meningioma Group: This group is based on the type of histopathology and MRI images that lead to a meningioma type brain tumor.
  After grouping, blood serum samples was collected to check the value of CRP, procalcitonin and NLR. The data were entered in a table and then compared with values from other types of brain tumors.
  Interventions: Diagnostic Test: Procalcitonin
- Glioma Group: This group is based on the type of histopathology and MRI images that lead to a glioma type brain tumor.
  After grouping, blood serum samples was collected to check the value of CRP, procalcitonin and NLR. The data were entered in a table and then compared with values from other types of brain tumors.
  Interventions: Diagnostic Test: Procalcitonin
- Brain Metastasis Group: This group is based on the type of histopathology and MRI images that lead to a metastasis brain tumor type After grouping, blood serum samples was collected to check the value of CRP, procalcitonin and NLR. The data were entered in a table and then compared with values from other types of brain tumors.
  Interventions: Diagnostic Test: Procalcitonin

INTERVENTIONS:
Diagnostic Test: Procalcitonin — Samples were categorized based on demographic data (age and gender), then the samples were categorized based on the type of brain tumor suffered. Once categorized, the levels of inflammatory markers was examined. Specimens were taken from the patient's peripheral blood examination and analyzed in laboratorium. The results of these examinations are grouped on a nominal scale, and analyzed statistically
  Other Names: C-Reactive Protein (CRP); Neutrophyl to Lymphocyte Ratio (NLR)

SUMMARY:
This study is a case controlled analytical study that analyzes the relationship between levels of inflammatory markers with the type of brain tumor. Samples of 35 people were then categorized according to the variables above and analyzing to measure its significance

DETAILED DESCRIPTION:
This study is a case controlled analytical study to find the relationship between levels of inflammatory markers in patients with brain tumors. Samples were collected from patients at Haji Adam Malik Hospital in Medan, then the patient's blood serum was taken to be checked for these variables. Sample collection began in March - September 2020. The sample obtained was 35 people who met the inclusion and exclusion criteria.

Inclusion criteria:

1. Willing to be a sample
2. Complete medical records
3. Head scan and head contrast MRI have been performed to confirm the patient's diagnosis with a brain tumor

Exclusion criteria:

1. The patient's age is over 70 years
2. Patients with high comorbidities such as kidney failure, heart disease, diabetes, and others
3. Patients with a history of brain tumor surgery or previous brain tumor treatment

Samples were categorized based on demographic data (age and gender), then the samples were categorized based on the type of brain tumor suffered. Once categorized, the levels of inflammatory markers was examined. Specimens were taken from the patient's peripheral blood examination and analyzed in laboratorium. The results of these examinations are grouped on a nominal scale, and analyzed statistically.

Based on this analysis, it will be determined whether there is a significant relationship between levels of inflammatory markers in the incidence of brain tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to be a sample
2. Complete medical records
3. Head scan and head contrast MRI have been performed to confirm the patient's diagnosis with a brain tumor

Exclusion Criteria:

1. The patient's age is over 70 years
2. Patients with high comorbidities such as kidney failure, heart disease, diabetes, and others
3. Patients with a history of brain tumor surgery or previous brain tumor treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Samples were collected from patients at Haji Adam Malik Hospital in Medan, Sample collection began in March - September 2020
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Value of Procalcitonin | February-April 2020
  Value of Procalcitonin in each group (Meningioma Group, Glioma Group and Brain metastasis group)
Value of C-Reactive Protein | April- June 2020
  Value of C-Reactive Protein in each group (Meningioma Group, Glioma Group and Brain metastasis group)
Value of Neutrophyl to Lymphocyte Ratio (NLR) | June- August 2020
  Value of NLR in each group (Meningioma Group, Glioma Group and Brain metastasis group)

SECONDARY OUTCOMES:
Demographic of samples | August- October 2020
  Demographic of each samples such as age, gender, Glassgow coma scale and Karnofsky score

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Universitas Sumatera Utara, Medan, North Sumatera, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Casado-Flores J, Blanco-Quiros A, Asensio J, Arranz E, Garrote JA, Nieto M. Serum procalcitonin in children with suspected sepsis: a comparison with C-reactive protein and neutrophil count. Pediatr Crit Care Med. 2003 Apr;4(2):190-5. doi: 10.1097/01.PCC.0000059420.15811.2D. PMID 12749651
- [Result] Quail DF, Joyce JA. Microenvironmental regulation of tumor progression and metastasis. Nat Med. 2013 Nov;19(11):1423-37. doi: 10.1038/nm.3394. PMID 24202395
- [Result] Engelhardt B, Vajkoczy P, Weller RO. The movers and shapers in immune privilege of the CNS. Nat Immunol. 2017 Feb;18(2):123-131. doi: 10.1038/ni.3666. Epub 2017 Jan 16. PMID 28092374
- [Result] Deutschman CS. Acute-phase responses and SIRS/MODS: the good, the bad, and the nebulous. Crit Care Med. 1998 Oct;26(10):1630-1. doi: 10.1097/00003246-199810000-00007. No abstract available. PMID 9781714
- [Result] Bambury RM, Teo MY, Power DG, Yusuf A, Murray S, Battley JE, Drake C, O'Dea P, Bermingham N, Keohane C, Grossman SA, Moylan EJ, O'Reilly S. The association of pre-treatment neutrophil to lymphocyte ratio with overall survival in patients with glioblastoma multiforme. J Neurooncol. 2013 Aug;114(1):149-54. doi: 10.1007/s11060-013-1164-9. Epub 2013 Jun 19. PMID 23780645
- [Result] Hatherill M, Tibby SM, Sykes K, Turner C, Murdoch IA. Diagnostic markers of infection: comparison of procalcitonin with C reactive protein and leucocyte count. Arch Dis Child. 1999 Nov;81(5):417-21. doi: 10.1136/adc.81.5.417. PMID 10519716
- [Result] Michelson N, Rincon-Torroella J, Quinones-Hinojosa A, Greenfield JP. Exploring the role of inflammation in the malignant transformation of low-grade gliomas. J Neuroimmunol. 2016 Aug 15;297:132-40. doi: 10.1016/j.jneuroim.2016.05.019. Epub 2016 May 25. PMID 27397086
- [Result] Sen E. Targeting inflammation-induced transcription factor activation: an open frontier for glioma therapy. Drug Discov Today. 2011 Dec;16(23-24):1044-51. doi: 10.1016/j.drudis.2011.09.003. Epub 2011 Sep 6. PMID 21920453
- [Result] Tracey KJ, Cerami A. Tumor necrosis factor, other cytokines and disease. Annu Rev Cell Biol. 1993;9:317-43. doi: 10.1146/annurev.cb.09.110193.001533. No abstract available. PMID 8280464
- [Result] D'Andrea A, Rengaraju M, Valiante NM, Chehimi J, Kubin M, Aste M, Chan SH, Kobayashi M, Young D, Nickbarg E, et al. Production of natural killer cell stimulatory factor (interleukin 12) by peripheral blood mononuclear cells. J Exp Med. 1992 Nov 1;176(5):1387-98. doi: 10.1084/jem.176.5.1387. PMID 1357073
- [Result] Voll RE, Herrmann M, Roth EA, Stach C, Kalden JR, Girkontaite I. Immunosuppressive effects of apoptotic cells. Nature. 1997 Nov 27;390(6658):350-1. doi: 10.1038/37022. No abstract available. PMID 9389474
- [Result] Balkwill F, Mantovani A. Inflammation and cancer: back to Virchow? Lancet. 2001 Feb 17;357(9255):539-45. doi: 10.1016/S0140-6736(00)04046-0. PMID 11229684
- [Result] Mantovani A, Allavena P, Sica A, Balkwill F. Cancer-related inflammation. Nature. 2008 Jul 24;454(7203):436-44. doi: 10.1038/nature07205. PMID 18650914
- [Result] Conti A, Guli C, La Torre D, Tomasello C, Angileri FF, Aguennouz M. Role of inflammation and oxidative stress mediators in gliomas. Cancers (Basel). 2010 Apr 26;2(2):693-712. doi: 10.3390/cancers2020693. PMID 24281089
- [Result] Faria SS, Fernandes PC Jr, Silva MJ, Lima VC, Fontes W, Freitas-Junior R, Eterovic AK, Forget P. The neutrophil-to-lymphocyte ratio: a narrative review. Ecancermedicalscience. 2016 Dec 12;10:702. doi: 10.3332/ecancer.2016.702. eCollection 2016. PMID 28105073
- [Result] Templeton AJ, Ace O, McNamara MG, Al-Mubarak M, Vera-Badillo FE, Hermanns T, Seruga B, Ocana A, Tannock IF, Amir E. Prognostic role of platelet to lymphocyte ratio in solid tumors: a systematic review and meta-analysis. Cancer Epidemiol Biomarkers Prev. 2014 Jul;23(7):1204-12. doi: 10.1158/1055-9965.EPI-14-0146. Epub 2014 May 3. PMID 24793958
- [Result] Zadora P, Dabrowski W, Czarko K, Smolen A, Kotlinska-Hasiec E, Wiorkowski K, Sikora A, Jarosz B, Kura K, Rola R, Trojanowski T. Preoperative neutrophil-lymphocyte count ratio helps predict the grade of glial tumor - a pilot study. Neurol Neurochir Pol. 2015;49(1):41-4. doi: 10.1016/j.pjnns.2014.12.006. Epub 2015 Jan 6. PMID 25666772